CLINICAL TRIAL: NCT02067130
Title: Utility of Transient Elastography (Fibroscan) in Estimating Hepatic Iron Concentration in Comparison to MRI in Patients With Transfusion Dependent Hemoglobinopathies
Brief Title: Utility of Fibroscan in Estimating Hepatic Iron Concentration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H13-02149
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Hereditary Anemias
Keywords: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fibroscan (Other): Subjects enrolled will undergo Fibroscan. It is an affordable and noninvasive tool for measuring liver stiffness as a predictor of liver fibrosis. Fibroscan reading will be collected at the Gastroenterologist's (Dr. Ko) outpatient clinic (Pacific Gastroenterology Associates) where a qualified research nurse/assistant will perform the scan under supervision of the physician. Anticipated timing of this procedure will be October to December 2013
  Interventions: Procedure: Fibroscan

INTERVENTIONS:
Procedure: Fibroscan — Transient elastography (Fibroscan®) is an affordable and noninvasive tool for measuring liver stiffness as a predictor of liver fibrosis. Since Fibroscan® measures liver's stiffness, its utility is not limited to fibrosis, and has been extended to other conditions that would increase the liver's stiffness, such as amyloidosis (Loustaud-Ratti et al. Amyloid 2011) and perhaps iron overload.

SUMMARY:
In patients with hereditary anemias (e.g. thalassemias), defective red blood cells are produced due to an error in the genes, or DNA, that provide the instructions for their synthesis. As a result, hereditary anemias are characterized by chronically low hemoglobin, which is contained inside red blood cells and carries oxygen throughout the body. In more severe cases, patients are dependent on frequent blood transfusions to replenish the hemoglobin.

The body has limited ability to get rid of excess iron. However, with repeated blood transfusions, the iron level in the body builds up because the red blood cells contain iron as heme. Over time, the high level of iron accumulates in organs such as the heart, liver, and pancreas causing heart problems, liver failure, and diabetes. As a result, patients who receive multiple blood transfusions need to be monitored for iron overload, and be started on medical therapy in a timely fashion to prevent organ damage.

Liver is usually the first and the most affected organ by iron accumulation, so knowledge of its iron concentration provides estimate of total body iron load. Liver biopsy is the gold standard in measuring the iron concentration in the liver, but it is invasive and cannot be performed on routine basis. MRI is another option that can assess liver iron concentration non-invasively, and is currently recommended for monitoring iron load on a yearly basis. However, MRI has a high cost and is not easily accessible in Canada. The investigators aim to determine if transient elastography (Fibroscan), which is a form of ultrasound that measures liver stiffness, can accurately assess liver iron concentration.

Hypothesis:

Fibroscan reading correlates with MRI and serum ferritin in estimating hepatic iron concentration.

DETAILED DESCRIPTION:
Inclusion criteria: All adult patients (age 19 or greater) with hereditary anemias requiring chronic blood transfusion at St. Paul's Hospital will be invited to participate in this study. The majority of patients will be β-Thalassemia Major. They will be given a pamphlet containing the details of the study and can contact the research assistant or clinic nurse for more information should they be interested.

Exclusion criteria: Patients with known Hepatitis B positive, known Hepatitis C positive, known HIV positive, known liver cirrhosis, known primary liver disease such as Wilson's disease and hereditary hemochromatosis are excluded from the study.

Written consent will be obtained from all participants by the clinic nurse/research assistant prior to enrollment.

Study procedures:

Data to be collected retrospectively from patient charts (St. Paul's Hospital's EMR/Sunrise Clinical Manager and paper chart) include: baseline demographic data (age, gender, hematological condition), medical comorbidities and complications related to iron overload (Diabetes, hypothyroidism, cardiomyopathy/arrhythmia and congestive heart failure, hypogonadotropic hypogonadism, osteopenia and osteoporosis syndrome..etc), current medications including use of iron chelators such as desferrioxamine, deferasirox, deferiprone or combination therapy, viral hepatitis status (B and C) and date of test, liver cirrhosis status (stage), liver biopsy result (iron concentration) and date of procedure. Patients with chronic transfusion requirement usually undergo annual MRI at the beginning of the year to estimate hepatic iron concentration as per standard practice. This year (2013), R2 MRI (FerriScan) will also be available for the first time to all patients in BC as part of routine monitoring for iron overload. Details/results from both techniques (i.e. same images collected in one scan, but analyzed differently using R2 and T2* algorithms) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age 19 or greater) with hereditary anemias requiring chronic blood transfusion at St. Paul's Hospital will be invited to participate in this study. The majority of patients will be β-Thalassemia Major.

Exclusion Criteria:

* Known Hepatitis B positive
* Known Hepatitis C positive
* Known HIV positive
* Known liver cirrhosis
* Known primary liver disease such as Wilson's disease and hereditary hemochromatosis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Fibroscan reading collected at the Gastroenterologist's outpatient clinic | 1 year
  Fibroscan results will be compared to that of T2* MRI, R2 MRI (FerriScan) and serum ferritin using linear regression models to determine if there is any correlation between FibroScan® results and liver iron concentration, which is indirectly measured with MRI and serum ferritin.

CONTACTS AND LOCATIONS:
Overall Officials: Hatoon Ezzat, MD, Principal Investigator — Department of Medicine, Division of Hematology St. Paul's Hospital, University of British Columbia; Hinhin Ko, MD, Principal Investigator — Department of Medicine, Division of Gastroenterology, St. Paul's Hospital, University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Shander A, Sazama K. Clinical consequences of iron overload from chronic red blood cell transfusions, its diagnosis, and its management by chelation therapy. Transfusion. 2010 May;50(5):1144-55. doi: 10.1111/j.1537-2995.2009.02551.x. Epub 2010 Jan 15. PMID 20088842
- [Background] Jung KS, Kim SU. Clinical applications of transient elastography. Clin Mol Hepatol. 2012 Jun;18(2):163-73. doi: 10.3350/cmh.2012.18.2.163. Epub 2012 Jun 26. PMID 22893866
- [Background] Loustaud-Ratti VR, Cypierre A, Rousseau A, Yagoubi F, Abraham J, Fauchais AL, Carrier P, Lefebvre A, Bordessoule D, Vidal E, Sautereau D, Jaccard A. Non-invasive detection of hepatic amyloidosis: FibroScan, a new tool. Amyloid. 2011 Mar;18(1):19-24. doi: 10.3109/13506129.2010.543443. Epub 2011 Jan 10. PMID 21219116
- [Background] Remacha A, Sanz C, Contreras E, De Heredia CD, Grifols JR, Lozano M, Nunez GM, Salinas R, Corral M, Villegas A; Spanish Society of Blood Transfusion; Spanish Society of Haematology and Haemotherapy. Guidelines on haemovigilance of post-transfusional iron overload. Blood Transfus. 2013 Jan;11(1):128-39. doi: 10.2450/2012.0114-11. Epub 2012 Jul 4. No abstract available. PMID 22790272
- [Background] Gandon Y, Olivie D, Guyader D, Aube C, Oberti F, Sebille V, Deugnier Y. Non-invasive assessment of hepatic iron stores by MRI. Lancet. 2004 Jan 31;363(9406):357-62. doi: 10.1016/S0140-6736(04)15436-6. PMID 15070565
- [Background] Hou P, Popat UR, Lindsay RJ, Jackson EF, Choi H. A practical approach for a wide range of liver iron quantitation using a magnetic resonance imaging technique. Radiol Res Pract. 2012;2012:207391. doi: 10.1155/2012/207391. Epub 2012 Dec 11. PMID 23365743
- [Background] Argyropoulou MI, Astrakas L. MRI evaluation of tissue iron burden in patients with beta-thalassaemia major. Pediatr Radiol. 2007 Dec;37(12):1191-200; quiz 1308-9. doi: 10.1007/s00247-007-0567-1. Epub 2007 Aug 21. PMID 17710390